CLINICAL TRIAL: NCT06929273
Title: A Phase 3, Open-label Extension Study to Assess the Long-term Safety of KarXT for the Treatment of Mania or Mania With Mixed Features in Bipolar-I Disorder (BALSAM-3)
Brief Title: A Study to Assess the Long-term Safety of KarXT for the Treatment of Manic Episodes in Bipolar-I Disorder (BALSAM-3)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CN012-0038; U1111-1316-9287 (Other: WHO); 2024-520259-26 (Other: EU CTR)
Record Dates: First submitted 2025-04-14; First posted 2025-04-16 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Bipolar Disorder Type I With Mania
Keywords: Bipolar-I disorder; Mania; Bipolar-I disorder with Mania
MeSH Terms: conditions — Mania | interventions — xanomeline; trospium chloride; Lithium; Valproic Acid; Lamotrigine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- KarXT or Adjuvant KarXT (Experimental)
  Interventions: Drug: KarXT; Drug: Lithium; Drug: Valproate; Drug: Lamotrigine

INTERVENTIONS:
Drug: KarXT — Specified dose on specified days
  Other Names: BMS-986510; Xanomeline and trospium chloride
Drug: Lithium — Therapeutic dose
Drug: Valproate — Therapeutic dose
Drug: Lamotrigine — Therapeutic dose

SUMMARY:
This is a phase 3, open-label extension study to assess the long-term safety of KarXT for the treatment of mania or mania with mixed features in Bipolar-I disorder (BP-I)

The primary objective of the study is to evaluate the long-term safety and tolerability of KarXT in the treatment of participants with mania or mania with mixed features associated with BP-I.

ELIGIBILITY:
Inclusion Criteria:

* Participants who participated in double-blind placebo-controlled study (CN0120036, CN0120037, or CN0120046):

  a. Participants must have completed treatment period of parent study.
* De novo participants who did not participate in double-blind placebo-controlled studies:

  1. Participants must have primary diagnosis of Bipolar-I disorder established by a comprehensive psychiatric evaluation based on DSM-5-TR criteria and confirmed by the Mini International Neuropsychiatric Interview (MINI, v7.0.2), with symptoms of mania or mixed mania.
  2. Participants must have Young Mania Rating Scale (YMRS) score of ≥ 14 at Screening and at baseline.
  3. Participants must have CGI-BP score of ≥ 3 at Screening and at baseline.
  4. Participants does not require hospitalization for acute mania.

Exclusion Criteria:

* Participants who participated in double-blind placebo-controlled study (CN0120036, CN0120037, or CN0120046):

  a. Discontinuation from any KarXT parent studies.
* De novo participants who did not participate in double-blind placebo-controlled studies:

  1. All participants with a risk for suicidal behavior at baseline as determined by Investigator's clinical assessment or history of suicidal behavior as assessed on C-SSRS.
  2. Participants must not have primary diagnosis of BP-I with rapid cycling (ie, ≥ 4 distinct mood episodes in one year).
  3. Participants must not have any primary DSM-5-TR disorder other than BP-I with mania or mania with mixed features within 12 months before Screening (confirmed using MINI version 7.0.2 at Screening), including BP-I with depression, (previous 3 months only), Bipolar-II disorder, major depressive disorder, borderline personality disorder, and primary psychotic disorder, with the exception of mild anxiety disorders.
  4. Individual has a DSM-5-TR diagnosis of moderate to severe substance use disorder (except tobacco use disorder) within the 12 months before Screening (confirmed using MINI version 7.0.2 at Screening), or current use as determined by urine toxicology screen or alcohol test.
  5. Participants must not have history of irritable bowel syndrome (with or without constipation) or serious constipation requiring treatment within the last 6 months.
  6. Participants must not have history or high risk of urinary retention, gastric retention, or untreated narrow-angle glaucoma.
  7. Other protocol-defined Inclusion/Exclusion criteria apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2025-07-18 (Actual); Primary Completion 2028-06-13 (Estimated); Study Completion 2028-06-13 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment emergent adverse events (TEAEs) | Up to week 54

SECONDARY OUTCOMES:
Number of participants with AEs of special interest (AESIs) | Up to week 54
Number of participants with serious AEs (SAEs) | Up to week 54
Number of participants with TEAEs leading to treatment discontinuation | Up to week 52
Number of participants with change in suicidal ideation as assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS) | Up to week 54
Change from baseline in Barnes Akathisia Rating Scale (BARS) score | Up to week 54
Change from baseline in Simpson Angus Scale (SAS) score | Up to week 54
Change from baseline in Abnormal Involuntary Movement Scale (AIMS) score | Up to week 54
Change from baseline in International Prostate Symptom Score (IPSS) | Up to week 54
  Only for males ≥ 45 years of age

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (166):
- United States (50):
  - Local Institution - 0120, Glendale, Arizona
  - Pillar Clinical Research - Richardson, Bentonville, Arkansas
  - Pillar Clinical Research- Little Rock, Little Rock, Arkansas
  - Woodland International Research Group, Little Rock, Arkansas
  - Woodland Research Northwest, Rogers, Arkansas
  - Advanced Research Center Inc., Anaheim, California
  - Clinical Innovations, Inc. dba CITrials, Bellflower, California
  - Local Institution - 0044, Cerritos, California
  - Local Institution - 0135, Chino, California
  - Proscience Research Group, Culver City, California
  - Collaborative Neuroscience Research, LLC, Garden Grove, California
  - Local Institution - 0137, La Habra, California
  - Catalina Research Institute, LLC, Montclair, California
  - NRC Research Institute, Orange, California
  - Clinical Innovations, Inc. dba CITrials, Riverside, California
  - Collaborative Neuroscience Research, LLC, Torrance, California
  - Local Institution - 0131, New Haven, Connecticut
  - Local Institution - 0133, Hallandale, Florida
  - Local Institution - 0026, Hialeah Gardens, Florida
  - Behavioral Clinical Research, Hollywood, Florida
  - Local Institution - 0053, Hollywood, Florida
  - LCC Medical Research Institute, Miami, Florida
  - Advanced Research Institute of Miami, Miami, Florida
  - Innovative Clinical Research, Inc., Miami Lakes, Florida
  - South Florida Research Phase I-IV, Miami Springs, Florida
  - Local Institution - 0045, St. Petersburg, Florida
  - Health Synergy Clinical Research, Stuart, Florida
  - Synexus Clinical Research US, Inc., Atlanta, Georgia
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - CenExel iResearch, LLC, Decatur, Georgia
  - CenExel iResearch, LLC, Savannah, Georgia
  - Local Institution - 0031, Chicago, Illinois
  - Pillar Clinical Research -Chicago, Chicago, Illinois
  - CBH Health, Gaithersburg, Maryland
  - Local Institution - 0029, Flowood, Mississippi
  - Arch Clinical Trials, St Louis, Missouri
  - Local Institution - 0121, North Las Vegas, Nevada
  - Local Institution - 0122, North Las Vegas, Nevada
  - Hassman Research Institute Marlton Site, Marlton, New Jersey
  - Local Institution - 0058, Marlton, New Jersey
  - Richmond Behavioral Associates, Staten Island, New York
  - Local Institution - 0124, Charlotte, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Neuro-Behavioral Clinical Research, North Canton, Ohio
  - Local Institution - 0134, Austin, Texas
  - InSite Clinical Research, DeSoto, Texas
  - Local Institution - 0046, Houston, Texas
  - Local Institution - 0138, Houston, Texas
  - Local Institution - 0036, Irving, Texas
  - Pillar Clinical Research - Richardson, Richardson, Texas
- Argentina (3):
  - Local Institution - 0128, ABB, Buenos Aires F.D.
  - Local Institution - 0127, Córdoba
  - Local Institution - 0126, Mendoza
- Australia (2):
  - Ramsay Clinic Northside, St Leonards, New South Wales
  - Ramsay Clinic New Farm, Brisbane, Queensland
- Bulgaria (5):
  - Center for Mental Health Prof. Dr. Ivan Temkov, Burgas
  - Local Institution - 0107, Novi Iskar
  - "University Multiprofile Hospital for Active Treatment - Dr. Georgi Stranski" EAD, Pleven
  - Local Institution - 0113, Sliven
  - Mental Health Center - Vratsa, Vratsa
- China (11):
  - Local Institution - 0177, Beijing, Beijing Municipality
  - Local Institution - 0174, Beijing, Beijing Municipality
  - Local Institution - 0175, Guangzhou, Guangdong
  - Local Institution - 0181, Baoding, Hebei
  - Local Institution - 0185, Shijiazhuang, Hebei
  - Local Institution - 0184, Changsha, Hunan
  - Local Institution - 0180, Nanjing, Jiangsu
  - Local Institution - 0176, Xi'an, Shaanxi
  - Local Institution - 0179, Chengdu, Sichuan
  - Local Institution - 0183, Tianjin, Tianjin Municipality
  - Local Institution - 0182, Ningbo, Zhejiang
- Croatia (5):
  - Local Institution - 0018, Zagreb, City of Zagreb
  - Local Institution - 0017, Zagreb
  - Local Institution - 0019, Zagreb
  - Local Institution - 0103, Zagreb
  - Local Institution - 0129, Zagreb
- Denmark (2):
  - Local Institution - 0154, Glostrup Municipality, Capital Region
  - Local Institution - 0153, Aalborg, North Denmark
- France (3):
  - Local Institution - 0170, Nice, Alpes-Maritimes
  - Local Institution - 0171, Clermont-Ferrand
  - Local Institution - 0172, Montpellier
- Hungary (3):
  - Petz Aladar Egyetemi Oktato Korhaz, Győr, Győr-Moson-Sopron
  - Local Institution - 0110, Budapest
  - Semmelweis Egyetem, Budapest
- India (10):
  - Local Institution - 0111, Vadodara, Gujarat
  - Local Institution - 0132, Belagavi, Karnataka
  - Local Institution - 0159, Mangalore, Karnataka
  - Local Institution - 0079, Kozhikode, Kerala
  - Local Institution - 0077, Ludhiana, Punjab
  - Local Institution - 0158, Madurai, Tamil Nadu
  - Local Institution - 0078, Hyderabad, Telangana
  - Local Institution - 0080, Hyderabad, Telangana
  - Local Institution - 0076, Kolkata, West Bengal
  - Local Institution - 0160, Kolkata, West Bengal
- Israel (8):
  - Shalvata Mental Health Center, Hod HaSharon, Central District
  - Local Institution - 0075, Ness Ziona, Central District
  - Local Institution - 0084, Petah Tikva, Central District
  - Sheba Medical Center, Ramat Gan, Central District
  - Be'er Sheva Mental Health Center, Beersheba, Southern District
  - Local Institution - 0173, Ashkelon
  - Local Institution - 0168, Jerusalem
  - Kfar Shaul Mental Health Center, Jerusalem
- Italy (5):
  - Local Institution - 0066, Milan, Lombardy
  - Local Institution - 0083, Pisa, Tuscany
  - Local Institution - 0065, Siena, Tuscany
  - Local Institution - 0070, Ancona
  - Local Institution - 0069, Genova
- Japan (24):
  - Hotei Hospital, Kōnan, Aichi-ken
  - Okehazama Hospital, Toyoake, Aichi-ken
  - National Kohnodai Medical Center., Ichikawa, Chiba
  - Local Institution - 0166, Iizuka, Fukuoka
  - Local Institution - 0063, Kitakyushu, Fukuoka
  - Obihiro Kosei Hospital, Obihiro, Hokkaido
  - Goryokai Medical Corporation - Goryokai Hospital, Sapporo, Hokkaido
  - Local Institution - 0165, Yokohama, Kanagawa
  - Kansai Medical University Medical Center, Moriguchi, Osaka
  - Local Institution - 0007, Sakai-shi, Osaka
  - Rainbow and Sea Hospital, Karatsu-shi, Saga-ken
  - Local Institution - 0016, Iruma, Saitama
  - Saitama Konan Hospital, Kumagaya, Saitama
  - Local Institution - 0163, Bunkyo-ku, Tokyo
  - Local Institution - 0164, Bunkyo-ku, Tokyo
  - National Center of Neurology and Psychiatry, Kodaira, Tokyo
  - Narimasu Kosei Hospital, tabashi City, Tokyo
  - Kuramitsu Hospital, Fukuoka
  - Local Institution - 0161, Kochi
  - Local Institution - 0004, Miyazaki
  - Osaka Metropolitan University Hospital, Osaka
  - Showa Medical University Karasuyama Hospital, Tokyo
  - Wakayama Medical University Hospital, Wakayama
  - Yamagata Sakuracho Hospital, Yamagata
- Local Institution - 0086, Auckland, New Zealand
- Poland (6):
  - Local Institution - 0088, Poznan, Greater Poland Voivodeship
  - Local Institution - 0092, Warsaw, Masovian Voivodeship
  - Local Institution - 0090, Bialystok, Podlaskie Voivodeship
  - Local Institution - 0093, Gdansk, Pomeranian Voivodeship
  - Local Institution - 0089, Rybnik, Silesian Voivodeship
  - Local Institution - 0091, Tuszyn, Łódź Voivodeship
- Romania (7):
  - Local Institution - 0095, Bucharest, București
  - Prof. Dr. Alexandru Obregia Psychiatry Hospital, Bucharest, București
  - Local Institution - 0167, Bucharest
  - Centrul de Evaluare și Tratament a Toxicodependenței pentru Tineri Sf.Stelian, Bucharest
  - Local Institution - 0094, Bucharest
  - Local Institution - 0097, Iași
  - Local Institution - 0100, Sanpetru /Brasov
- Slovakia (3):
  - Local Institution - 0118, Košice, Košice Region
  - Local Institution - 0119, Košice, Košice Region
  - Local Institution - 0117, Vranov nad Topľou, Presov
- Spain (3):
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona [Barcelona]
  - Osi Bilbao-Basurto, Bilbao, Basque Country
  - Hospital Clínic de Barcelona, Barcelona, Catalunya [Cataluña]
- Sweden (3):
  - Nacka Local Hospital, Nacka, Stockholms Län [se-01]
  - Local Institution - 0112, Uppsala, Uppsala Län [se-03]
  - Local Institution - 0116, Gothenburg, Västra Götalands Län [se-14]
- Ukraine (12):
  - Local Institution - 0152, Smila, Cherkasy Oblast
  - Local Institution - 0149, Dnipro, Dnipropetrovsk Oblast
  - Local Institution - 0142, Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - Local Institution - 0146, Skarzhyntsi, Khmelnytskyi Oblast
  - Local Institution - 0143, Hlevakha, Kyiv Oblast
  - Local Institution - 0150, Kyiv, Kyivska Oblast
  - Local Institution - 0147, Lviv, Lviv Oblast
  - Local Institution - 0145, Oleksandrivka, Odesa Oblast
  - Local Institution - 0141, Poltava, Poltava Oblast
  - Local Institution - 0148, Vinnytsia, Vinnytsia Oblast
  - Local Institution - 0151, Kropyvnytskyi
  - Local Institution - 0144, Odesa

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT06929273.html